CLINICAL TRIAL: NCT00653939
Title: A Phase II Study to Assess the Safety and Efficacy of the Combination of Carboplatin, Paclitaxel, and Bevacizumab ± Combretastatin A4 Phosphate (CA4P) Followed by Bevacizumab ± CA4P in Subjects With Chemotherapy Naïve Stage IIIB/IV Non-Squamous Cell Histology Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Safety and Efficacy Study of Carboplatin, Paclitaxel, Bevacizumab and CA4P in Non-Small Cell Lung Cancer
Acronym: FALCON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXC401-216
Record Dates: First submitted 2008-03-18; First posted 2008-04-07 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Tumors
Keywords: non-small cell lung cancer; non-small cell lung carcinoma; neoplasms, lung; lung cancer; tumors; NSCLC
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — fosbretabulin; Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Chemotherapy+Bevacizumab (Active Comparator): Carboplatin (AUC 6), paclitaxel (200 mg/m2), and bevacizumab (15 mg/kg)administered intravenously on Day 1 of a 21-day cycle for up to six treatment cycles. After 6 cycles, subjects who have not progressed may continue to receive bevacizumab (15 mg/kg) alone on Day 1 every 3 weeks until progression or until 12 months from randomization.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab
- Arm 2: Active Comparator+Fosbretabulin (Experimental): Carboplatin (AUC 6), paclitaxel (200 mg/m2), and bevacizumab (15 mg/kg), administered intravenously Day 1 of a 21-day cycle and fosbretabulin (60 mg/m2) on Days 7, 14, and 21 for up to six treatment cycles. After 6 cycles, subjects who have not progressed may continue to receive bevacizumab (15 mg/kg) on Day 1 and fosbretabulin on Days 1, 7 and 14 every 3 weeks until progression or until 12 months from randomization.
  Interventions: Drug: Fosbretabulin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Fosbretabulin — Arm 2 only: Fosbretabulin (60 mg/m2) on Days 7,14 and 21 for 6 cycles.
  Other Names: Combretastatin A4 Phosphate; Zybrestat; CA4P
  Arms: Arm 2: Active Comparator+Fosbretabulin
Drug: Carboplatin — Chemotherapy: Carboplatin (AUC 6) on Day 1 of each 21 day cycle for 6 cycles.
  Other Names: Paraplatin
Drug: Paclitaxel — Chemotherapy: Paclitaxel (20 mg/m2) on Day 1 of each 21-day cycle for 6 cycles.
  Other Names: Taxol
Drug: Bevacizumab — Bevacizumab (15 mg/kg) on Day 1 of each 21-day cycle for 6 cycles.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of combretastatin A4 phosphate (CA4P), also known as fosbretabulin, in combination with bevacizumab (Avastin), carboplatin and paclitaxel in patients with chemotherapy naïve non-small cell lung cancer (NSCLC). This is a randomized parallel arm study. All participants will receive carboplatin, paclitaxel and bevacizumab, and half will additionally receive CA4P. Patients who complete the first 6 cycles of therapy and have not experienced disease progression will receive maintenance therapy with bevacizumab alone or with bevacizumab plus CA4P.

The rationale for this study is the potential additive or synergistic actions of vascular disrupting agents like CA4P with anti-angiogenic agents like bevacizumab.

DETAILED DESCRIPTION:
Lung cancer has become the leading cause of cancer death in both men and women in the US and Europe, accounting for 29% of all cancer deaths. Non-Small Cell Lung cancer (NSCLC) accounts for approximately 80% of all lung cancer cases. Currently, no curative treatment is available for advanced stages of the disease (stages III and IV), which comprise the majority of cases. Treatment with the combination of carboplatin and paclitaxel has been shown to be effective and well tolerated in advanced stage NSCLC. Targeted therapies, such as bevacizumab, often act synergistically with chemotherapy. Bevacizumab inhibits vascular endothelial growth factor (VEGF), necessary for endothelial cell proliferation and new blood vessel formation. CA4P targets existing abnormal vasculature of tumors, impeding tumor blood flow and leading to extensive tumor cell death as a consequence of oxygen and nutrient deprivation.

This study will compare the effect of CA4P when combined with chemotherapy and bevacizumab on progression free survival (PFS) to PFS after chemotherapy and bevacizumab alone.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Stage IIIB NSCLC with malignant pleural effusion, or Stage IV disease
* Measurable disease on CT scan (by the Response Evaluation Criteria in Solid Tumors [RECIST] criteria)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1 (which means able to independently care for self and to perform light work) .
* Adequate blood counts
* Adequate liver and kidney function
* Subjects or their legal representatives must be able to read, understand and provide written informed consent to participate in the trial.

Exclusion Criteria:

* Predominant Squamous Cell NSCLC histology.
* History of treatment for NSCLC with chemotherapy, biological therapy, immunotherapy (surgery or radiation therapy are accepted)
* Brain (CNS) metastasis by head CT scan or MRI
* Subjects with history of prior malignancy except for curatively treated basal cell carcinoma of the skin; cervical intra-epithelial neoplasia; or localized prostate cancer with a current prostate specific antigen (PSA) of < 4.0 mg/dL. Subjects with other curatively treated malignancies who have no evidence of metastatic disease and >2 year disease free interval may be entered after discussion with the Medical Monitor.
* History of bleeding disorders, particularly coughing up ≥ ½ teaspoon bright red blood during the last 3 months
* Certain cardiac disorders such as recent myocardial infarction (MI), severe congestive heart failure, certain types of abnormal cardiac rhythm
* Uncontrolled high blood pressure despite medications
* Uncontrolled, clinically significant active infection.
* Known HIV
* Known hypersensitivity to any of the components of CA4P, paclitaxel, carboplatin, bevacizumab, or radiologic contrast dyes.

Details of the above and additional inclusion and exclusion criteria can be discussed with an investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Balkissoon, MD, FACS, Study Director — Mateon Therapeutics
Locations (15):
- United States (15):
  - Southbay Oncology Hematology, Campbell, California
  - Pacific Coast Hematology and Oncology Medical Group, Fountain Valley, California
  - UCLA Division of Hematology and Oncology, Los Angeles, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Gabrail Cancer Center, Canton, Ohio
  - The Mark H. Zangmeister Center, Columbus, Ohio
  - Signal Point Clinical Research, Middletown, Ohio
  - Blueridge Cancer Care, Salem, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - Mary Babb Randolph Cancer Center-Clinical Trials Unit, Morgantown, West Virginia

REFERENCES:
- [Background] Lin CM, Singh SB, Chu PS, Dempcy RO, Schmidt JM, Pettit GR, Hamel E. Interactions of tubulin with potent natural and synthetic analogs of the antimitotic agent combretastatin: a structure-activity study. Mol Pharmacol. 1988 Aug;34(2):200-8. PMID 3412321
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Monestiroli S, Mancuso P, Burlini A, Pruneri G, Dell'Agnola C, Gobbi A, Martinelli G, Bertolini F. Kinetics and viability of circulating endothelial cells as surrogate angiogenesis marker in an animal model of human lymphoma. Cancer Res. 2001 Jun 1;61(11):4341-4. PMID 11389057
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Chaplin DJ, Pettit GR, Hill SA. Anti-vascular approaches to solid tumour therapy: evaluation of combretastatin A4 phosphate. Anticancer Res. 1999 Jan-Feb;19(1A):189-95. PMID 10226542
- [Background] Siemann DW, Mercer E, Lepler S, Rojiani AM. Vascular targeting agents enhance chemotherapeutic agent activities in solid tumor therapy. Int J Cancer. 2002 May 1;99(1):1-6. doi: 10.1002/ijc.10316. PMID 11948484
- [Background] Shaked Y, Ciarrocchi A, Franco M, Lee CR, Man S, Cheung AM, Hicklin DJ, Chaplin D, Foster FS, Benezra R, Kerbel RS. Therapy-induced acute recruitment of circulating endothelial progenitor cells to tumors. Science. 2006 Sep 22;313(5794):1785-7. doi: 10.1126/science.1127592. PMID 16990548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Started | 31 (2 patients randomized did not receive treatment due to brain metastasis or consent withdrawal.) | 32 (1 patient randomized did not receive treatment due to acute renal failure.)
Completed | 19 | 17
Not Completed | 12 | 15
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 4 | 0
Not completed — Disease Progression | 2 | 3
Not completed — Other | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Chemotherapy+Bevacizumab: Carboplatin (AUC 6), paclitaxel (200 mg/m2), and bevacizumab (15 mg/kg) administered intravenously on Day 1 of a 21-day cycle for up to six treatment cycles. After 6 cycles, subjects who have not progressed may continue to receive bevacizumab (15 mg/kg) alone on Day 1 every 3 weeks until progression or until 12 months from randomization.
  Carboplatin: Chemotherapy: Carboplatin (AUC 6) on Day 1 of each 21 day cycle for 6 cycles.
  Paclitaxel: Chemotherapy: Paclitaxel (20 mg/m2) on Day 1 of each 21-day cycle for 6 cycles.
  Bevacizumab: Bevacizumab (15 mg/kg) on Day 1 of each 21-day cycle for 6 cycles.
- Arm 2: Active Comparator+Fosbretabulin: Carboplatin (AUC 6), paclitaxel (200 mg/m2), and bevacizumab (15 mg/kg), administered intravenously Day 1 of a 21-day cycle and fosbretabulin (60 mg/m2) on Days 7, 14, and 21 for up to six treatment cycles. After 6 cycles, subjects who have not progressed may continue to receive bevacizumab (15 mg/kg) on Day 1 and fosbretabulin on Days 1, 7 and 14 every 3 weeks until progression or until 12 months from randomization.
  Fosbretabulin: Arm 2 only: Fosbretabulin (60 mg/m2) on Days 7, 14 and 21 for 6 cycles.
  Carboplatin: Chemotherapy: Carboplatin (AUC 6) on Day 1 of each 21 day cycle for 6 cycles.
  Paclitaxel: Chemotherapy: Paclitaxel (20 mg/m2) on Day 1 of each 21-day cycle for 6 cycles.
  Bevacizumab: Bevacizumab (15 mg/kg) on Day 1 of each 21-day cycle for 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.5) | 61.0 (9.4) | 62.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 12 | 19 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 27 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: participants]
  0 - Fully active | 16 | 16 | 32
  1 - Restricted in physically strenuous activity | 13 | 15 | 28
Surgery Performed [Number; unit: participants]
  Yes | 5 | 4 | 9
  No | 24 | 27 | 51
Prior Surgery Due to NSCLC [Number; unit: participants]
  Yes | 3 | 2 | 5
  No | 26 | 29 | 55
Subject Given Radiation Therapy [Number; unit: participants]
  Yes | 5 | 4 | 9
  No | 23 | 27 | 50
  Information Missing | 1 | 0 | 1
Prior Radiation Due to NSCLC [Number; unit: participants]
  Yes | 4 | 4 | 8
  No | 25 | 27 | 52
Stage of Disease at Study Entry [Number; unit: participants]
  IIIB | 4 | 2 | 6
  IV | 25 | 29 | 54

OUTCOME MEASURES:

1. Secondary Outcome: Best Overall Tumor Response Rate (RR) in the Intent-to-Treat Population
Description: Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 for target lesions (assessed by MRI or CT scan): Complete Response (CR) is defined as the disappearance of all target lesions, Partial Response (PR) is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, Progressive Disease is defined as at least 20% increase in the sum of the longest diameter of target lesions, Stable Disease (SD) is defined as neither shrinkage to qualify for a PR or increase to qualify for a PD.
Time Frame: Six 21-day cycles
Population: Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Number analyzed (Participants) | 31 | 32
participants
  Complete Response | 0 | 0
  Partial Response | 11 | 18
  Stable Disease | 13 | 8
  Progressive Disease | 3 | 1
  Unknown | 4 | 5

2. Secondary Outcome: Overall Survival (OS) Using a Multivariate Cox Regression Model in the Intent-to-Treat Population
Time Frame: Until death or lost to follow-up, up to 12 months since randomization
Population: Intent-to-Treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Number analyzed (Participants) | 31 | 32
Months | 16.2 [9.9 to 17.7] | 13.6 [8.6 to 17.8]

3. Primary Outcome: Progression Free Survival (PFS) in the Intent-to-Treat Population
Description: Progression was defined using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0. Based on 20% increase of the longest diameter of target lesions or appearance of one or more new non-target lesions or/and progression of non-target lesions since the treatment started.
Time Frame: Six 21-day cycles
Population: Intent-to-Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Number analyzed (Participants) | 31 | 32
months | 9.3 [4.4 to 11.5] | 8.6 [5.0 to 10.2]

4. Secondary Outcome: Chemistry NCI-CTCAE Toxicity Grade of 3 or 4 (Safety Population)
Time Frame: Days 1 (pretreatment) per 21-day Cycle (6 Cycles)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Number analyzed (Participants) | 29 | 31
participants
  ALT - Grade 3 | 1 | 1
  ALT - Grade 4 | 0 | 0
  AST - Grade 3 | 0 | 1
  AST - Grade 4 | 0 | 0
  ALP - Grade 3 | 0 | 0
  ALP - Grade 4 | 0 | 0
  Total Bilirubin - Grade 3 | 0 | 0
  Total Bilirubin - Grade 4 | 0 | 0
  Glucose - Grade 3 | 0 | 0
  Glucose - Grade 4 | 1 | 0
  Creatinine - Grade 3 | 0 | 0
  Creatinine - Grade 4 | 1 | 1
  Calcium - Grade 3 | 3 | 0
  Calcium - Grade 4 | 1 | 1
  Magnesium - Grade 3 | 2 | 1
  Magnesium - Grade 4 | 2 | 1
  Phosphorus - Grade 3 | 0 | 1
  Phosphorus - Grade 4 | 0 | 0
  Potassium - Grade 3 | 5 | 0
  Potassium - Grade 4 | 1 | 0
  Sodium - Grade 3 | 5 | 2
  Sodium - Grade 4 | 0 | 0

5. Secondary Outcome: Hematology NCI-CTCAE Grade 3 or 4 (Safety Population)
Time Frame: Days 1 (pretreatment), 7, 14, and 21 per 21-day Cycle (6 Cycles)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Number analyzed (Participants) | 29 | 31
participants
  Hemoglobin - Grade 3 | 7 | 0
  Hemoglobin - Grade 4 | 4 | 1
  White Blood Cell - Grade 3 | 14 | 12
  White Blood Cell - Grade 4 | 2 | 1
  Absolute Neutrophils - Grade 3 | 4 | 5
  Absolute Neutrophils - Grade 4 | 20 | 20
  Platelets - Grade 3 | 3 | 5
  Platelets - Grade 4 | 6 | 3

6. Secondary Outcome: Coagulation NCI-CTCAE Grade 3 or 4 (Safety Population)
Time Frame: Day 1 (pretreatment) per 21-day Cycle (6 Cycles)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Number analyzed (Participants) | 29 | 31
participants
  INR - Grade 3 | 2 | 3
  INR - Grade 4 | 0 | 0
  PTT - Grade 3 | 3 | 5
  PTT - Grade 4 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1: Chemotherapy+Bevacizumab | Arm 2: Active Comparator+Fosbretabulin
Serious Adverse Events (participants affected / at risk) | 16/29 | 16/31
Other Adverse Events (participants affected / at risk) | 29/29 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Chemotherapy+Bevacizumab (N=29) | Arm 2: Active Comparator+Fosbretabulin (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 2
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Disease Progression (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Infusion Site Thrombosis (General disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Arthritis Infective (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Lung Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pseudomonal Bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cerbral Infarction (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epixtaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Repiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Chemotherapy+Bevacizumab (N=29) | Arm 2: Active Comparator+Fosbretabulin (N=31)
Neutropenia (Blood and lymphatic system disorders) | 14 | 25
Anaemia (Blood and lymphatic system disorders) | 20 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 13
Leukopenia (Blood and lymphatic system disorders) | 7 | 14
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 20 | 13
Diarrhoea (Gastrointestinal disorders) | 17 | 11
Constipation (Gastrointestinal disorders) | 11 | 11
Vomiting (Gastrointestinal disorders) | 11 | 7
Abdominal Pain (Gastrointestinal disorders) | 5 | 5
Stomatitis (Gastrointestinal disorders) | 3 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 1
Gingival Bleeding (Gastrointestinal disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 4 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Oral Pain (Gastrointestinal disorders) | 1 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 25 | 18
Pyrexia (General disorders) | 10 | 6
Oedema peripheral (General disorders) | 6 | 8
Asthenia (General disorders) | 6 | 4
Chest Discomfort (General disorders) | 2 | 5
Chills (General disorders) | 3 | 2
Gait Disturbance (General disorders) | 2 | 3
Non-cardiac Chest Pain (General disorders) | 2 | 3
Mucosal Inflammation (General disorders) | 1 | 3
Pain (General disorders) | 3 | 1
Chest Pain (General disorders) | 1 | 2
Infusion Site Pain (General disorders) | 0 | 3
Adverse Drug Reaction (General disorders) | 0 | 2
Neuropathy (Nervous system disorders) | 19 | 15
Headache (Nervous system disorders) | 12 | 4
Dizziness (Nervous system disorders) | 9 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 6
Dysgeusia (Nervous system disorders) | 3 | 3
Burning Sensation (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 2 | 2
Amnesia (Nervous system disorders) | 0 | 2
Balance Disorder (Nervous system disorders) | 0 | 2
Memory Impairment (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 3
Anorexia (Metabolism and nutrition disorders) | 9 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 6
Dehydration (Metabolism and nutrition disorders) | 8 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pharyngolarygeal Pain (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 10 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 9
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 13
Rash (Skin and subcutaneous tissue disorders) | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Upper Respiratory Tract Infections (Infections and infestations) | 4 | 5
Urinary Tract Infection (Infections and infestations) | 6 | 3
Bronchitis (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 4 | 0
Catheter Site Infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 1
Fungal Infection (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 1 | 2
Oral Candidiasis (Infections and infestations) | 2 | 0
Tooth Infection (Infections and infestations) | 0 | 2
Hypertension (Vascular disorders) | 13 | 17
Hypotension (Vascular disorders) | 7 | 1
Flushing (Vascular disorders) | 1 | 4
Orthostatic Hypotension (Vascular disorders) | 5 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 3
Weight Decreased (Investigations) | 8 | 3
Alanine Aminotransferase Increased (Investigations) | 3 | 1
Breath Sounds Abnormal (Investigations) | 1 | 3
Gamma-glutamyltransferase Increased (Investigations) | 2 | 2
Blood Chloride Decreased (Investigations) | 0 | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 2
Blood Urea Increased (Investigations) | 2 | 0
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 2
Oxygen Saturation Decreased (Investigations) | 2 | 0
Prothrombin Time Prolonged (Investigations) | 0 | 2
Insomnia (Psychiatric disorders) | 5 | 7
Depression (Psychiatric disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 3 | 2
Confusional State (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 3 | 8
Bradycardia (Cardiac disorders) | 0 | 4
Angina Pectoris (Cardiac disorders) | 2 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 3
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 5 | 3
Haematuria (Renal and urinary disorders) | 2 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 1
Vision Blurred (Eye disorders) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1
Ear Pain (Ear and labyrinth disorders) | 2 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 1 | 2
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Endocrine Disorders (Endocrine disorders) | 2 | 1
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No